CLINICAL TRIAL: NCT05236036
Title: A Phase 1/1b Adaptive Dose Escalation Study of Mycophenolate Mofetil (MMF) in Combination With Standard of Care for Patients With Glioblastoma
Brief Title: Mycophenolate Mofetil in Combination With Standard of Care for the Treatment of Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NU 21C01; NCI-2021-12424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00215766; NU 21C01 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Astrocytoma; Glioblastoma; Glioblastoma, IDH-Wildtype; MGMT-Unmethylated Glioblastoma; Recurrent Glioblastoma
MeSH Terms: conditions — Astrocytoma; Glioblastoma | interventions — Mycophenolic Acid; Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (TMZ, MMF) (Experimental): Patients who have already undergone surgery or biopsy followed by chemoradiation receive TMZ PO QD on days 1-5 of each cycle and MMF PO BID. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mycophenolate Mofetil; Other: Quality-of-Life Assessment; Drug: Temozolomide
- Group 2 (TMZ, MMF, radiation therapy) (Experimental): Patients with unmethylated glioblastoma who have already undergone surgery or biopsy receive TMZ PO QD on days 1-5 of each cycle and MMF PO BID. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Starting at the same time as TMZ and MMF administration, patients also receive radiation therapy daily, 5 days per week, for 6 weeks.
  Interventions: Drug: Mycophenolate Mofetil; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Temozolomide
- Group 3 (TMZ, MMF, radiation therapy) (Experimental): Patients who have already undergone surgery or biopsy receive TMZ PO QD on days 1-5 of each cycle and MMF PO BID. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Starting at the same time as TMZ and MMF administration, patients also receive radiation therapy daily, 5 days per week, for 6 weeks.
  Interventions: Drug: Mycophenolate Mofetil; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Temozolomide
- Group S (pre-surgical MMF, TMZ) (Experimental): Patients planning to undergo surgery receive MMF PO BID and TMZ PO QD for 5 days prior to surgery in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mycophenolate Mofetil; Other: Quality-of-Life Assessment; Drug: Temozolomide

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Given PO
  Other Names: CellCept; MMF
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Receive radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Group 2 (TMZ, MMF, radiation therapy); Group 3 (TMZ, MMF, radiation therapy)
Drug: Temozolomide — Given Orally (PO)
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I/Ib trial tests the safety, side effects, and best dose of mycophenolate mofetil in combination with temozolomide and/or radiation therapy (standard of care) in treating patients with glioblastoma. Mycophenolate mofetil is an immunosuppressant drug that is typically used to prevent organ rejection in transplant recipients. However, mycophenolate mofetil may also help chemotherapy with temozolomide work better by making tumor cells more sensitive to the drug. The purpose of this trial is to determine if mycophenolate mofetil combined with temozolomide can stop glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the recommended phase 2 dose (RP2D) for mycophenolate mofetil (MMF) in combination with radiation therapy as well as in combination with temozolomide (TMZ).

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of mycophenolate mofetil (MMF) in combination with temozolomide (TMZ).

II. To estimate progression free survival (PFS) per Response Assessment in Neuro-Oncology Criteria (RANO).

III. To estimate overall survival (OS). IV. To estimate the overall response rate (ORR) per RANO criteria. V. To evaluate quality of life per Functional Assessment of Cancer Therapy Scale-Brain (FACT-Br) for patients treated with mycophenolate mofetil and/or temozolomide.

EXPLORATORY OBJECTIVES:

I. To investigate the relationship between the molecular signature of individual glioblastoma multiforme (GBM) with clinical outcome, by measuring levels of serum mycophenolic acid in patient's plasma post MMF administration.

Ia. Perform molecular characterization of all GBM tissues by ribonucleic acid sequencing (RNAseq) analysis.

Ib. Perform bulk metabolomics for GBM tissue. Ic. Measure plasma and serum concentration of mycophenolic acid, the MMF's primary active metabolite, during and after combination therapy.

Id. Measure IMPDH activity assay in patients' peripheral blood mononuclear cells (PBMCs) as well as in GBM tissue.

OUTLINE: This is a dose-escalation study of MMF (Part 1), followed by a dose-expansion study (Part 2).

PART 1: Patients are assigned to 1 of 3 groups.

GROUP 1: Patients who have already undergone surgery or biopsy followed by chemoradiation receive TMZ orally (PO) once daily (QD) on days 1-5 of each cycle and MMF PO twice daily (BID). Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

GROUP 2: Patients with unmethylated glioblastoma who have already undergone surgery or biopsy receive TMZ PO QD on days 1-5 of each cycle and MMF PO BID. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Starting at the same time as TMZ and MMF administration, patients also receive radiation therapy daily, 5 days per week, for 6 weeks.

GROUP S: Patients planning to undergo surgery receive MMF PO BID and TMZ PO QD for 5 days prior to surgery in the absence of disease progression or unacceptable toxicity.

PART 2: Patients are assigned to Group 3.

GROUP 3: Patients who have already undergone surgery or biopsy receive TMZ PO QD on days 1-5 of each cycle and MMF PO BID. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Starting at the same time as TMZ and MMF administration, patients also receive radiation therapy daily, 5 days per week, for 6 weeks.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* GROUPS 1-3: Histologically confirmed glioblastoma (GBM), IDH wild-type (by immunohistochemistry [IHC] R132H negative [neg] or sequencing). Astrocytoma with molecular features of GBM are eligible.
* GROUPS 1-3: Newly diagnosed glioblastoma and:

  * Group 1: Received surgical resection or biopsy followed by chemoradiation;
  * Group 2: Received surgical resection or biopsy only and have documented unmethylated glioblastoma (may have been done at an outside facility);
  * Group 3: Received surgical resection or biopsy only
* GROUP S: Newly suspected glioblastoma or recurrent glioblastoma, and scheduled to undergo a standard of care surgical resection or biopsy.
* Stable or decreasing dose of corticosteroids equivalent to =< 8 mg dexamethasone daily, for >= 7 days prior to registration.

  * Note: There are no restrictions on steroid use on study
* Patients must be age >= 18 years.
* Patients must exhibit a Karnofsky performance status >= 70.
* Leukocytes (white blood cells [WBC]) >= 3,000/mcL (within 14 days prior to study registration)
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 14 days prior to study registration)
* Hemoglobin (Hgb) >= 8 g/dL (within 14 days prior to study registration) (transfusion may be used for eligibility if >= 7 days)
* Platelets (PLT) >= 100,000/mcL (within 14 days prior to study registration) (transfusion or growth factor may be used for eligibility if >= 7 days).
* Total bilirubin =< 2x institutional upper limit of normal (ULN) (within 14 days prior to study registration)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/Alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN (within 14 days prior to study registration)
* Creatinine =< 1.5 x Institutional ULN (within 14 days prior to study registration)
* International normalized ratio (INR) =< 1.5 x ULN (within 14 days prior to study registration)
* Prothrombin time (PT)/Partial thromboplastin Time (PTT) =< 1.5 x ULN (within 14 days prior to study registration)
* Females of child-bearing potential (FOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent, for the duration of study participation, and for 3 months following completion of therapy. Should a female patient become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception from time of informed consent, for the duration of study participation, and 4 months after completion of administration.

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test within 14 days prior to registration on study.
* Patient or their legally authorized representative must provide written, signed, and dated informed consent prior to study registration. Patient or their legally authorized representative (LAR) must have the ability to understand and the willingness to sign a written informed consent document. The patient or their LAR must be willing and able to comply with the protocol for the duration of the study.

  * NOTE: no study-specific screening procedures may be performed until written consent has been obtained.

Exclusion Criteria:

* Patients who are receiving any other investigational agents.

  * Exception: COVID-19 vaccine and treatment is allowed
* Patient who have a prior or concurrent malignancy that may interfere with study treatment or safety.

  * NOTE: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible. Per principal investigator (PI) discretion
* Patients who have a history of allergic reactions attributed to compounds of similar chemical composition to temozolomide or mycophenolate mofetil.
* Patients with spinal cord and diffuse leptomeningeal disease GBM
* Patients requiring live vaccinations within 2 weeks of initiation of MMF and/or TMZ therapy. Consider completion of vaccination with live vaccines prior to starting immunosuppressive therapy, as indicated.
* Patients on viral-vector based therapy due to increased risk for disseminated herpetic infection.
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Have uncontrolled epilepsy
  * Have an uncontrolled intercurrent illness
  * Concurrent malignancy (outside of glioblastoma) that requires tumor directed treatment
  * Known deficiency of hypoxanthine-guanin-phosphoribosyltransferase (HGPRT) deficiency, e.g. Lesch-Nyhan- oder Kelley-Seegmiller-Syndrome.
  * Known concurrent shingles, herpes, CMV (cytomegalovirus) infection
  * Known concurrent opportunistic fungal infection
  * Known concurrent or history of unexplained opportunistic infection
  * Known immunodeficiency that could lead to opportunistic infections
  * Psychiatric illness/social situations that would limit compliance with study requirements. Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints.
* Female patients who are pregnant or nursing. Pregnant women are excluded from this study because temozolomide is an alkylating agent with potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with temozolomide, breastfeeding should be discontinued if the mother is treated with temozolomide.
* Patients who are unable to swallow oral medication or have problems/ diseases that affect absorption of oral medication.
* Patients with a known history of human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV).

  * Note: Temozolomide and mycophenolate mofetil are immunosuppressive agents. Patients with a known history of HIV, HBV, and HCV, and unexplained opportunistic infections are not eligible due to safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2029-01-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) for mycophenolate mofetil (MMF) (Group 1) | Up to completion of first cycle of treatment + 7 days (1 cycle = 28 days)
  Will be based on treatment-emergent and drug related toxicity of grade >= 3 during the first cycle of treatment. MTD indicates maximum tolerated dose for dose limiting toxicity (DLT). DLT is defined as side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment. Recommended phase 2 dose (RP2D) is the highest dose of a drug or treatment that does not cause unacceptable side effects. For the purposes of this study, RP2D is interchangeable with MTD. DLTs and Adverse Events (AEs) will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v). 5.0.
MTD/RP2D for MMF (Group 2) | Up to 6 weeks + 7 days
  Will be based on treatment-emergent and drug related toxicity of grade >= 3 during focal radiation treatment. MTD indicates maximum tolerated dose for DLT. DLT is defined as side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment. RP2D is the highest dose of a drug or treatment that does not cause unacceptable side effects. For the purposes of this study, RP2D is interchangeable with MTD. DLTs and AEs will be assessed by CTCAE v.5.0.

SECONDARY OUTCOMES:
Frequency of adverse events | Up to 30 days after completion of study treatment
  The occurrence of toxicity (including [AEs] and serious adverse events [SAEs]), and the number of patients who discontinue treatment due to toxicity, as assessed by CTCAE v. 5.0. This endpoint will collect and report the frequency of adverse events by type, severity (grade), timing, and attribution to MMF, according the National Cancer Institute (NCI)-CTCAE v. 5.0.
Progression Free Survival (PFS) | From baseline until the patient experiences disease progression, initiates subsequent anti-cancer therapy, completes study participation, or experiences death from any cause (whichever is sooner), assessed up to 18 months
  Progression will be determined by clinical progression or by radiographic imaging as assessed by Response Assessment in Neuro-Oncology Criteria (RANO). If disease progression or death from any cause is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the PFS will be censored as the last available disease assessment. Kaplan-Meier curves will be plot. Log-rank test will be used to compare it with historical standard care control in literature.
Overall survival (OS) | From time of diagnosis until the patient initiates subsequent anti-cancer therapy, completes study participation, or experiences death from any cause (whichever is sooner), assessed up to 18 months
  If death from any cause is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the OS will be censored as the last available follow-up. will be described by Kaplan-Meier curve. The median and corresponding 95% confidence interval will also be estimated.
Overall response rate (ORR) | From baseline, the patient experiences disease progression, the patient initiates subsequent anti-cancer therapy, or the patient completes study participation (whichever occurs first), assessed up to 18 months
  Overall response rate will be assessed by RANO criteria. To determine the ORR, this endpoint will calculate the proportion of treated patients who experience an overall response (complete response [CR] or partial response [PR] per RANO criteria). The date of first response for either CR or PR will be used for the calculation of ORR. Will be estimated using the expansion cohort, along with its 95% confidence interval.
Quality of life (QOL) | Up to 6 cycles (1 cycle = 28 days)
  The quality of life indicated by FACT-Br will be evaluated by estimating its mean, standard deviation and 95% confidence interval using the expansion cohort. Patients who received at least 1 dose of temozolomide (TMZ) and/or MMF, and completed at least baseline and cycle 2 day 1 (C2D1) FACT-Br QOL (for Groups 1-3) will be evaluable for this secondary endpoint.

OTHER OUTCOMES:
Mycophenolic acid levels | Days 1, 3 and 7 post-MMF administration for cycles 1 and 2
  Will measure in patients' plasma by using the Food and Drug Administration (FDA)-approved protocol Analytical Chemistry Division at the Illinois Institute of Technology Research Institute.
XMP concentration | Up to 6 cycles (1 cycle = 28 days)
  Will utilize an established clinical protocol and a highly sensitive liquid chromatography-mass spectrometry method in peripheral blood mononuclear cells (PBMCs) isolated from glioblastoma patients receiving MMF in combination with TMZ in order to determine IMPDH activity. This is a clinically validated protocol in which the analytical methods yielded acceptable within samples and within individual variability. Peripheral blood samples taken at baseline and day 1 of each adjuvant TMZ+MMF cycle will be used to test this.

CONTACTS AND LOCATIONS:
Overall Officials: Priya U Kumthekar, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois
  - Northwestern Medicine Warrenville, Warrenville, Illinois